CLINICAL TRIAL: NCT02161523
Title: The Impact of Lung Cancer-derived Fibroblasts on Mast Cells Activation
Status: Completed | Type: Observational
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 0059-14-MMC; 0059-14-MMC (Other: Meir Medical Center)
Record Dates: First submitted 2014-06-10; First posted 2014-06-11 (Estimated); Last update posted 2018-03-22 (Actual); Status verified 2018-03

CONDITIONS: Lung Cancer
Keywords: mast cells, lung cancer, cancer associated fibroblasts (CAF)
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Biopsy from lung tissue

SUMMARY:
In addition to their role in allergic inflammation, mast cells are often found at the site of tumors. They have been attributed both to pro- and anti-tumorigenic roles depending on the tumor type. Secretion of mast cell mediators such as histamine, tryptase, fibroblast growth factor (b-FGF), vascular endothelial growth factor (VEGF) and interleukin-8 (IL-8) can enhance tumor growth and angiogenesis while TNF-a and heparin act as tumor suppressors.

The non-small cell lung cancer constitutes the majority of cases of lung cancer. In lung cancer, mast cell numbers correlate with tumor angiogenesis and poor prognosis.

In this work, we are interested to determine the factors in lung cancer microenvironment that attribute to mast cell activation. Beside the tumor cells themselves, the cancer microenvironment includes other cells such as fibroblasts. The fibroblasts arising from tumor stroma, called cancer-associated fibroblasts (CAFs), undergo activation, and have different feature compared to normal fibroblasts (NFs). In this work we are interested to determine whether CAF cells derived from lung tumors, together with the lung cancer cells, or microvesicles-derived from these cells, are able to stimulate mast cells to degranulate and/ or to release various cytokines and chemokines.

For this propose, during surgery of patients with lung cancer, we will take unnecessary sample from the cancer and from normal area for purification of CAF or normal fibroblast cells. Those cells will be co-cultured with both lung cancer cell line (A-549) or microvesicles-derived from these cells, and human mast cell line (LAD2). Supernatants will be collected for determine degranulation and cytokine release from these mast cells.

ELIGIBILITY:
Inclusion Criteria:

Patient with non small cell lung carcinoma

Exclusion Criteria:

none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patient with non small cell lung carcinoma that need a surgery without connection to this experiment
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2014-07-01 (Actual); Primary Completion 2015-06-01 (Actual); Study Completion 2015-06-01 (Actual)

PRIMARY OUTCOMES:
Measuring the levels of b-hexosaminidase (marker for mast cells degranulation ) and the cytokines levels | 1-2 weeks